CLINICAL TRIAL: NCT01024985
Title: Evaluation of Macular and Retinal Nerve Fiber Layer Thickness Measurements for Detection of Neural Loss in Multiple Sclerosis and Neuromyelitis Optica Using High Resolution Optical Coherence Tomography.
Brief Title: Evaluation of Neural Loss in Multiple Sclerosis and Neuromyelitis Optica Using High Resolution Oct
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: mario luiz ribeiro monteiro, university of sao paulo
Other Study IDs: 0190/09
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica
Keywords: optic neuritis; longitudinally extensive transverse myelitis; retinal nerve fiber layer; macular thickness
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Optic Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- multiple sclerosis
- neuromyelitis optica
- controls

SUMMARY:
The purpose of this study is to determine the ability of STRATUS OCT and high resolution OCT to detect and to quantify the neural loss in multiple sclerosis and neuromyelitis optica and its subtypes.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of multiple sclerosis or neuromyelitis optica
* age between 15 and 60 years
* BCVA better than 20/400
* no optic neuritis crisis in the last 6 months

Exclusion Criteria:

* diagnosis of glaucoma, opacities or disc anomalies
* diagnosis of macular disease
* disc swelling at fundoscopy

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients of ophthalmology and/or neurology departments of hopital das clinicas of medical school of university of sao paulo
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Das Clinicas Medical School of University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Hokazono K, Raza AS, Oyamada MK, Hood DC, Monteiro ML. Pattern electroretinogram in neuromyelitis optica and multiple sclerosis with or without optic neuritis and its correlation with FD-OCT and perimetry. Doc Ophthalmol. 2013 Dec;127(3):201-15. doi: 10.1007/s10633-013-9401-2. Epub 2013 Jul 30. PMID 23892551
- [Derived] Monteiro ML, Fernandes DB, Apostolos-Pereira SL, Callegaro D. Quantification of retinal neural loss in patients with neuromyelitis optica and multiple sclerosis with or without optic neuritis using Fourier-domain optical coherence tomography. Invest Ophthalmol Vis Sci. 2012 Jun 26;53(7):3959-66. doi: 10.1167/iovs.11-9324. PMID 22589446